CLINICAL TRIAL: NCT06253975
Title: A Randomized, Controlled, Multicenter Study of Human Adipose Tissue Derived Extracellular Vesicles Promoting Wound Healing
Brief Title: Randomized, Controlled, Multicenter Study of Extracellular Vesicles From Human Adipose Tissue Promoting Wound Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Drkailiu-RCT
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Wound Heal
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT-EV group (Experimental)
  Interventions: Biological: adipose tissue derived extracellular vesicles (AT-EVs)
- HA group (Placebo Comparator)
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Biological: adipose tissue derived extracellular vesicles (AT-EVs) — Extracellular vesicles from patient's adipose tissue together with HA
  Arms: AT-EV group
Drug: Hyaluronic acid — Use HA only as a placebo
  Arms: HA group

SUMMARY:
By randomly assigning study subjects into groups, interventions with adipose tissue-derived extracellular vesicles (AT-EVs) and placebos are conducted to evaluate whether AT-EVs can promote effective healing of recalcitrant wounds.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 69 years old, regardless of gender 2. Full-layer skin ulcers on various parts of the body, lasting from 4 weeks to 1 year

  1. If the wound is post-amputation, the time from surgery must be >30 days;
  2. If there is >1 wound surface, the maximum wound surface is selected as the research target; 3. At the beginning of the induction period, the wound size after debridement was ≥1 and ≤20 cm2; 4.Texas classification 1A, 1B, 1C, 1D, 2A, 2B, 2C or 2D; 5. Ankle-brachial index ≥0.7, including percutaneous oxygen pressure (TcPO2) ≥30 mm Hg and cutaneous perfusion pressure ≥30 mm Hg; 6. Revascularization procedures or vascular surgery that are not scheduled in the past or the next 30 days; 7. The subject and family members are willing and able to comply with all prescribed care and medical requirements; 8. The subject has a reasonable expectation of completing the study; 9. The subject completed the 2-week induction period and the wound was reduced by 30%

Exclusion Criteria:

* 1. The subject has signs of gangrene in any part of the trunk and limbs; 2. A written diagnosis of osteomyelitis in any part of the affected limb; 3. Bone tissue at the wound site of the subject is exposed; 4. Poor blood glucose control in subjects: HbA1c>12% (108 mmol/mol); 5. Subjects are receiving renal dialysis treatment or creatinine >2.5mg/dl (221mmol/L); 6. The subject has obvious immune deficiency; 7. The subject has suspected tumor or is receiving tumor treatment; 8. Subject has used steroids or immunosuppressants in the past 3 months or is expected to use them during the study; 9. Subjects received growth factor therapy, autologous platelet-rich plasma gel, double-layer cell therapy, dermal substitute, extracellular matrix, etc., during the screening period; 10. The subject has participated in another research device, drug, or biological trial within the past 30 days; 11. The wound shows serious clinical symptoms of infection, requiring hospitalization or immediate surgical treatment; 12. The subject has developed deep vein thrombosis within the past 30 days; 13. The subject is pregnant or breastfeeding; 14. The subject has serious mental illness and psychological disorder; 15. The subject was judged unfit for the test by the attending physician.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of wound healing in each group at 10 weeks | 10 weeks
  The percentage of wound healing in each group at 10 weeks was calculated as: (initial wound area - wound area at 10 weeks of treatment)/initial wound area ×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Liu, M.D., Ph.D., Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai 9th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No